CLINICAL TRIAL: NCT02296385
Title: Response to PUFA Intervention According to PPAR Genotypes
Brief Title: Genotype-related Effects of PUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11.16.NRC
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supplementation (Experimental): Supplementation
  Interventions: Dietary Supplement: Triple Strength Fish Oil

INTERVENTIONS:
Dietary Supplement: Triple Strength Fish Oil — Triple Strength Fish Oil

SUMMARY:
To assess the bioefficacy of omega-3 fatty acids (provided by intake of fish oil supplements) depending on genotype of relevant factors in lipid metabolism

DETAILED DESCRIPTION:
To assess the bioefficacy of omega-3 fatty acids (provided by intake of fish oil supplements) depending on genotype of relevant factors in lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult between 18 and 40 years of age
* BMI between 18.5 and 30 kg/m2
* Sedentary to moderate physical activity habits

Exclusion Criteria:

* Concomitant treatment: Consumption of dietary supplements or any medication that can affect the study outcomes
* Actively smoking
* Suspected abuse of alcohol or illicit drugs
* Significant illness within the two weeks prior to study start or any active systemic infection or medical condition that may require treatment during the study
* Known or suspected medical condition related to coagulation
* Subject who cannot be expected to comply with the study procedures
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to beginning of this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in triglyceride levels in plasma | Baseline and 6 weeks intervention

SECONDARY OUTCOMES:
Assess bioefficacy of EPA and DHA supplementation | Baseline and 6 weeks intervention
  The bioefficacy will be evaluated by characterizing and measuring the effects on lipid metabolism, glucose metabolism and insulin resistance, and inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elizabeth Tejero Barrera, PhD, Principal Investigator — Instituto Nacional de Medicina Genomica

REFERENCES:
- [Derived] Binia A, Vargas-Martinez C, Ancira-Moreno M, Gosoniu LM, Montoliu I, Gamez-Valdez E, Soria-Contreras DC, Angeles-Quezada A, Gonzalez-Alberto R, Fernandez S, Martinez-Conde D, Hernandez-Moran B, Ramirez-Solano M, Perez-Ortega C, Rodriguez-Carmona Y, Castan I, Rubio-Aliaga I, Vadillo-Ortega F, Marquez-Velasco R, Bojalil R, Lopez-Alvarenga JC, Valet P, Kussmann M, Silva-Zolezzi I, Tejero ME. Improvement of cardiometabolic markers after fish oil intervention in young Mexican adults and the role of PPARalpha L162V and PPARgamma2 P12A. J Nutr Biochem. 2017 May;43:98-106. doi: 10.1016/j.jnutbio.2017.02.002. Epub 2017 Feb 10. PMID 28282585